CLINICAL TRIAL: NCT05305885
Title: An Open-label, Randomized, Multicenter Trial of Intrathecal-pemetrexed Combined With Concurrent Involved-field Radiotherapy and Intrathecal-pemetrexed Alone in Patients With Leptomeningeal Metastasis From Solid Tumors
Brief Title: Intra-pemetrexed Alone or Combined With Concurrent Radiotherapy for Leptomeningeal Metastasis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Hospital of Jilin University (Other)
Collaborators: The Second Hospital of Hebei Medical University (Other); Second Affiliated Hospital of Guangzhou Medical University (Other); Affiliated Hospital of Guangdong Medical University (Other); Guangdong 999 Brain Hospital (Other); Wuxi People's Hospital (Other); Huizhou Third People's Hospital, Guangzhou Medical University (Other); Panjin Liaoyou Gem Flower Hospital (Unknown)
Responsible Party: Principal Investigator, Zhenyu Pan, Professor, The First Hospital of Jilin University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PMRT
Record Dates: First submitted 2022-03-14; First posted 2022-03-31 (Actual); Last update posted 2022-09-30 (Actual); Status verified 2022-09

CONDITIONS: Leptomeningeal Metastasis
Keywords: Leptomeningeal metastasis; Malignant solid tumors; Pemetrexed; Intrathecal chemotherapy; Radiotherapy
MeSH Terms: conditions — Meningeal Carcinomatosis | interventions — Pemetrexed; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Intrathecal administration, intraventricular administration or via lumbar puncture, pemetrexed plus dexamethasone, first induction intra-cerebrospinal fluid chemotherapy twice per week for 2 weeks, then once per week for 4 times, 6 weeks in total. Concurrent radiotherapy consisted of fractionated, conformal radiation given at a daily dose of 2 Gy. The planning volume consisted of sites of symptomatic disease, bulky disease observed on MRI, including the whole brain and basis cranii received 40 Gy in 20 fractions, 4 weeks in total, and/or segment of spinal canal received 40 Gy.
  Interventions: Drug: Pemetrexed; Radiation: Radiotherapy
- Group 2 (Experimental): Intrathecal administration, intraventricular administration or via lumbar puncture, pemetrexed plus dexamethasone, first induction intra-cerebrospinal fluid chemotherapy twice per week for 2 weeks, then once per week for 4 times, 6 weeks in total.
  Interventions: Drug: Pemetrexed

INTERVENTIONS:
Drug: Pemetrexed — Intrathecal administration, intraventricular administration or via lumbar puncture, pemetrexed plus dexamethasone, first induction intra-cerebrospinal fluid chemotherapy twice per week for 2 weeks, then once per week for 4 times, 6 weeks in total.
Radiation: Radiotherapy — Concurrent radiotherapy consisted of fractionated, conformal radiation given at a daily dose of 2 Gy. The planning volume consisted of sites of symptomatic disease, bulky disease observed on MRI, including the whole brain and basis cranii received 40 Gy in 20 fractions, 4 weeks in total, and/or segment of spinal canal received 40 Gy.
  Arms: Group 1

SUMMARY:
Intrathecal chemotherapy is one of the mainstay treatment options for leptomeningeal metastases. Owing to the limited number of agents available for intrathecal chemotherapy, it is crucial to find a novel agent with efficacy and safety. In our phase 1 study, intrathecal pemetrexed showed controllable toxicities and potential promising efficacy for refractory leptomeningeal metastases from non-small-cell lung cancer patients. In our further study, intrathecal pemetrexed combined with involved-field radiation therapy was administered as the first-line intrathecal chemotherapy for leptomeningeal metastases from solid tumors. In this study, intrathecal pemetrexed combined with involved-field radiation therapy showed feasibility and controllable adverse events. It has been proved that pemetrexed as a novel intrathecal drug exhibited promising antitumor effects in cerebrospinal fluid. Moreover, the concomitant therapeutic modality is an optimal treatment option for leptomeningeal metastases from solid tumors.

Central nervous system radiotherapy is a part of the specific treatment of leptomeningeal metastases. Radiotherapy has been proved to improve neurologic function and control of parenchymal brain metastases in leptomeningeal metastases treatment. Additionally, radiotherapy is revealed to improve the efficacy and attenuate toxicity of intrathecal chemotherapy as a result of normal cerebrospinal fluid reestablishing. However, it is still controversial whether radiotherapy can improve the overall survival. We conduct this study to further demonstrate the efficacy and safety of intrathecal pemetrexed administration for patients with leptomeningeal metastases from solid tumors by multicenter study. Furthermore, the study of effective treatment modality is of great significance. The safety and antitumor activity of intrathecal pemetrexed combined with involved-field radiation therapy and intrathecal pemetrexed alone were also compared to confirm an optimized therapeutic regimen.

DETAILED DESCRIPTION:
In this randomized, open-label, multicenter clinical trial, we aim to compare the efficacy and safety of intrathecal pemetrexed combined with concomitant involved-field radiation therapy and intrathecal pemetrexed alone for leptomeningeal metastasis patients from solid tumor. Patients were randomly divided into two arms willing to receive involved-field radiation therapy combined with concurrent intrathecal pemetrexed and intrathecal pemetrexed alone, respectively. In concomitant therapy group, participants received induction intrathecal pemetrexed first. Then concomitant intrathecal pemetrexed and involved-field radiation therapy were given. In intrathecal pemetrexed alone group, participants received induction intrathecal pemetrexed and consolidation intrathecal pemetrexed. Pemetrexed was administrated by intrathecal injection via intraventricular administration or lumbar puncture. Induction intrathecal pemetrexed was given twice per week for 2 weeks to all participants first. Then consolidation/concomitant intrathecal pemetrexed was given once per week for 4 weeks. Involved-field radiation therapy was administrated with a total dose of 40 Gy in 20 fractions for 4 weeks to the concomitant therapy group participants. Primary endpoints were clinical response and treatment-related adverse events. Secondary endpoints were overall survival and neurological progression-free survival.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a confirmed or probable diagnosis of leptomeningeal metastasis according to European Association of Neuro-Oncology-European Society for Medical Oncology (EANO-ESMO) guidelines；Patients who have been definitely diagnosed as leptomeningeal metastasis according to cerebrospinal fluid cytology, or patients who got the clinical diagnosis by combining with neuroimaging, history of cancer, clinical manifestation, cerebrospinal fluid examination, etc.
2. Participants with histologically or cytologically confirmed disease from solid tumors;
3. No history of whole brain radiotherapy;
4. Normal liver and kidney function; WBC≥4000/mm3, Plt≥100000/mm3.

Exclusion Criteria:

1. Patients with primary tumor of hematological tumors or primary central germ cell tumors;
2. Patients administrated with new molecular targeted therapy which is effective for leptomeningeal metastasis in 2 weeks;
3. Patients with hydrocephalus or other factors suggestive of cerebrospinal fluid circulation obstruction;
4. Patients with severe encephalopathy, grade 3 leukoencephalopathy, Glasgow Coma Scale less than 8 score;
5. Patients with extensive and lethal systemic diseases with few treatment options;
6. Patients with poor compliance, or for other reasons, the researchers considered unsuitable to participate in this clinical study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-08-19 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Clinical response rate | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 6 months.
  The response assessment in neuro-oncology criteria (RANO) proposal for response criteria of leptomeningeal metastasis was used to assess the clinical response in this study.
Incidence of treatment-related adverse events | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 6 months.
  The incidence of treatment-related adverse events were measured for determining tolerability and safety. Adverse events (AEs) are evaluated according to the Common Terminology Criteria for Adverse Events (CTCAE, version 4.03). Events of grade 3-5 are defined as moderate and severe adverse events.

SECONDARY OUTCOMES:
Overall survival | From the enrollment of this study until date of death from any cause, whichever came first, or the last follow-up (at least 7 months).
  Survival time was recorded since the date of patient enrollment. All patients were followed up until death or the end of the study.
Neurological progression-free survival (NPFS) | From date of randomization until the date of first documented neurological progression or date of death from any cause, whichever came first, assessed up to 6 months.
  NPFS was defined as time from the start of treatment until neurological progression or death. The neurological progression was determined based on the RANO proposal evaluation criteria which have been established and published on Neuro Oncol.

CONTACTS AND LOCATIONS:
Overall Officials: Zhenyu Pan, PhD., Principal Investigator — The First Hospital of Jilin University
Locations (1):
- The First Hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data that underlie results in a publication will be available to other researchers.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Starting 6 months after publication.
Access Criteria: Individual participant data will be public accessable via contacting with principal investigator by email within 6 months after the trial complete.

REFERENCES:
- [Background] Pan Z, Yang G, He H, Cui J, Li W, Yuan T, Chen K, Jiang T, Gao P, Sun Y, Cong X, Li Z, Wang Y, Pang X, Song Y, Zhao G. Intrathecal pemetrexed combined with involved-field radiotherapy as a first-line intra-CSF therapy for leptomeningeal metastases from solid tumors: a phase I/II study. Ther Adv Med Oncol. 2020 Jul 17;12:1758835920937953. doi: 10.1177/1758835920937953. eCollection 2020. PMID 32733606
- [Background] Pan Z, Yang G, He H, Gao P, Jiang T, Chen Y, Zhao G. Identification of Cerebrospinal Fluid MicroRNAs Associated With Leptomeningeal Metastasis From Lung Adenocarcinoma. Front Oncol. 2020 Apr 3;10:387. doi: 10.3389/fonc.2020.00387. eCollection 2020. PMID 32328453
- [Background] Pan Z, Yang G, Cui J, Li W, Li Y, Gao P, Jiang T, Sun Y, Dong L, Song Y, Zhao G. A Pilot Phase 1 Study of Intrathecal Pemetrexed for Refractory Leptomeningeal Metastases From Non-small-cell Lung Cancer. Front Oncol. 2019 Aug 30;9:838. doi: 10.3389/fonc.2019.00838. eCollection 2019. PMID 31544065